CLINICAL TRIAL: NCT03860220
Title: A Multi-center, Randomized, Parallel Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Triple Therapy of Telmisartan/Amlodipine/Rosuvastatin in Patients With Dyslipidemia and Hypertension
Brief Title: The Efficacy and Safety of Triple Therapy of Telmisartan/Amlodipine/Rosuvastatin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hyo-Soo Kim (Other)
Responsible Party: Sponsor-Investigator, Hyo-Soo Kim, Director, Coronary Intervention & Transcatheter Aortic Valve Implantation, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAROS
Record Dates: First submitted 2019-01-14; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — amlodipine, atorvastatin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEWSTATIN TS (Active Comparator): Triple therapy (Telmisartan + Amlodipine + Rosuvastatin 40/5/10mg)
  Interventions: Drug: NEWSTATIN TS
- CADUET (Placebo Comparator): Dual therapy (Amlodipine + Atorvastatin 5/10mg)
  Interventions: Drug: CADUET

INTERVENTIONS:
Drug: NEWSTATIN TS — Wash out/run in period with Amlodipine 5mg for 6 weeks and then treatment with triple therapy (Newstatin TS 40/5/10mg) ; 1 tab qd for 8 weeks
  Other Names: Newstatin TS 40/5/10mg
  Arms: NEWSTATIN TS
Drug: CADUET — Wash out/run in period with Amlodipine 5mg for 6 weeks and then treatment with dual therapy (Caduet 5/10mg) ; 1 tab qd for 8 weeks
  Other Names: Caduet 5/10mg
  Arms: CADUET

SUMMARY:
The goal of this study was to assess the efficacy and safety of FDC therapy with triple therapy of Telmisartan 40 mg/Amlodipine 5 mg/Rosuvastatin 10mg in Korean patients with both hypertension and dyslipidemia.

DETAILED DESCRIPTION:
Patients were randomly assigned to 2 groups: (1) Triple therapy (40mg of telmisartan and 5mg of amlodipine and 10mg of rosuvastatin); (2) Dual therapy (5mg of amlodipine and 10mg of atorvastatin). After 8 weeks of treatment, the change in mean sitting systolic blood pressure (MSSBP) and the percent change in LDL-C between 2 group, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 145 mmHg ≤ msSBP ≤ 190 mmHg
* Triglycerides < 500 mg/dL
* LDL-C ≤ 250 mg/dL

Exclusion Criteria:

* sSBP ≥ 20mmHg and sDBP ≥ 10mmHg
* symptomatic orthostatic hypotension and secondary/iatrogenic hypertension and dyslipidemia
* history of moderate to severe cerebral ischemia, cerebral hemorrhage, transient ischemic attack, myocardial infarction, or unstable angina in the past 6 months; severe heart failure (New York Heart Association functional class III and IV)
* hypersensitivity to telmisartan or rosuvastatin
* history of angioedema after treatment with angiotensin-converting enzyme inhibitors or ARBs; creatinine phosphokinase levels ≥3 times the upper limit of normal
* estimated glomerular filtration rate ≤30 mL/min; aspartate aminotransferase and alanine aminotransferase levels ≥3 times the upper limit of normal
* potassium levels >5.5 mmol/L; or any diseases that could affect the results of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent changes in mean sitting systolic blood pressure (MSSBP) | 8 weeks
  Percent changes in MSSBP from baseline after 8 weeks of treatment
Percent changes in LDL-C | 8 weeks
  Percent changes in LDL-C from baseline after 8 weeks of treatment

SECONDARY OUTCOMES:
Percent changes in LDL-C | 4 weeks
  Percent changes in LDL-C from baseline after 4 weeks of treatment
Percent changes in TC | 4, 8weeks
  Percent changes in TC from baseline after 4 and 8 weeks of treatment
Percent changes in TG | 4, 8weeks
  Percent changes in TG from baseline after 4 and 8 weeks of treatment
Percent changes in HDL-C | 4, 8weeks
  Percent changes in HDL-C from baseline after 4 and 8 weeks of treatment
Percent changes in Non-HDL-C | 4, 8weeks
  Percent changes in Non-HDL-C from baseline after 4 and 8 weeks of treatement
Percent changes in Apo B | 4, 8weeks
  Percent changes in Apo B from baseline after 4 and 8 weeks of treatment
Percent changes in Apo A-I | 4, 8weeks
  Percent changes in Apo A-I from baseline after 4 and 8 weeks of treatment
Percent changes in LDL-C/HDL-C ratio | 4, 8weeks
  Percent changes in LDL-C/HDL-C from baseline after 4 and 8 weeks of treatement
Percent changes in Apo B/Apo A-I ratio | 4, 8weeks
  Percent changes in Apo B/Apo A-I from baseline after 4 and 8 weeks of treatment
Percent changes in hs-CRP | 4, 8weeks
  Percent changes in hs-CRP from baseline after 4 and 8 weeks of treatment
The percentage of patients achieving treatment goal for blood pressure and LDL-C | 8 weeks
  The percentage of patients achieving treatment goal for blood pressure and LDL-C
Changes in mean sitting systolic/diastolic blood pressure | 4, 8weeks
  Changes in mean sitting systolic/diastolic blood pressure after 4 and 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park S, Hwang D, Kang J, Han JK, Yang HM, Park KW, Kang HJ, Koo BK, Cho JM, Cho BR, Ahn SG, Kang SM, Sung JH, Kim U, Lee N, Kim HS. Efficacy and Safety of Triple Therapy of Telmisartan/Amlodipine/Rosuvastatin in Patients with Dyslipidemia and Hypertension: A Multicenter Randomized Clinical Trial. Curr Ther Res Clin Exp. 2024 Feb 1;100:100735. doi: 10.1016/j.curtheres.2024.100735. eCollection 2024. PMID 38380420